CLINICAL TRIAL: NCT01149044
Title: TOTAL Trial: A Randomized Trial of Routine Aspiration ThrOmbecTomy With PCI Versus PCI ALone in Patients With STEMI Undergoing Primary PCI
Brief Title: A Trial of Routine Aspiration Thrombectomy With Percutaneous Coronary Intervention (PCI) Versus PCI Alone in Patients With ST-Segment Elevation Myocardial Infarction (STEMI) Undergoing Primary PCI
Acronym: TOTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Sanjit S. Jolly, MD MSc, FRCP(C), Interventional Cardiologist, Assistant Professor, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOTAL Trial
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Percutaneous Coronary Intervention
Keywords: Acute Coronary Syndrome; PCI; Percutaneous Coronary Intervention; STEMI; Thrombectomy
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Upfront Thrombectomy followed by PCI (Active Comparator): Upfront manual aspiration thrombectomy followed by PCI
  Interventions: Procedure: Percutaneous Coronary Intervention with or without manual aspiration thrombectomy
- PCI Alone (Active Comparator): PCI without upfront manual aspiration thrombectomy
  Interventions: Procedure: Percutaneous Coronary Intervention with or without manual aspiration thrombectomy

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention with or without manual aspiration thrombectomy

SUMMARY:
This is an international, randomized, controlled, parallel group study in which patients with ST-Segment Elevation Myocardial Infarction (STEMI) will be allocated to one of the following: Manual aspiration thrombectomy with Percutaneous Coronary Intervention (PCI) or PCI alone.

DETAILED DESCRIPTION:
The hypothesis for TOTAL is that the routine use of manual aspiration thrombectomy with an aspiration catheter (Export®) with PCI compared to PCI alone will reduce the incidence of cardiovascular death, recurrent myocardial infarction, cardiogenic shock, or new or worsening NYHA Class IV heart failure (HF) at 180 days in patients with STEMI undergoing primary PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with:

   * Symptoms of myocardial ischemia lasting for ≥ 30 minutes AND
   * Definite ECG changes indicating STEMI: ST elevation of greater than 0.1 mV in two contiguous limb leads or 0.2 mV in two contiguous precordial leads
2. Referred for primary PCI
3. Randomized within 12 hours of symptoms onset and prior to diagnostic angiography
4. Informed consent

Exclusion Criteria:

1. Age ≤ 18 years
2. Prior coronary artery bypass surgery (CABG)
3. Life expectancy less than six months due to non-cardiac condition
4. Treatment with fibrinolytic therapy for qualifying index STEMI event

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10732 (Actual)
Dates: Start 2010-08; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The first occurrence of cardiovascular death, recurrent myocardial infarction, cardiogenic shock, or new or worsening NYHA Class IV heart failure | up to 180 days

SECONDARY OUTCOMES:
Stroke | up to 30 days
Key Net Benefit Outcome: The first occurence of CV death, MI, stroke, cardiogenic shock or new or worsening NHYA Class IV heart failure | up to 1 year
Cardiovascular Mortality | up to 180 days
Key Secondary Efficacy Outcome: The first occurence of cardiovascular death, myocardial infarction, cardiogenic shock, new or worsening NYHA class IV heart failure, stent thrombosis and target vessel revascularization | up to 180 days

OTHER OUTCOMES:
Primary outcome at 30 days and 1 year | up to 1 year
Components of primary outcome and secondary outcomes | up to 1 year
  CV death, MI, cardiogenic shock, new or worsening class IV heart failure, stroke, stent thrombosis, target vessel revascularization assessed separately at 30 days, 180 days and one year
All-cause mortality | up to 1 year
  All-cause mortality at 30 days, 180 days and 1 year
Composite of CV death, MI, cardiogenic shock, or new or worsening NYHA class IV heart failure at 30 days, 180 days | up to 180 days
  Composite of cardiovascular death, myocardial infarction, cardiogenic shock, or new or worsening NYHA class IV heart failure at 30 days, 180 days
TIMI flow rates, no reflow | up to 1 year
Stent thrombosis | up to 1 year
Distal embolization | up to 1 year
Left main thrombus as a complication of the PCI procedure | up to 1 year
Target Vessel dissection | up to 1 year
Left main dissection | up to 1 year
Major Bleeding | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit S. Jolly, MD, MSc, FRCP, Principal Investigator — Hamilton Health Sciences Corporation; Vladimir Džavík, MD, FRCPC, Principal Investigator — Peter Munk Cardiac Centre, University Health Network
Locations (87):
- United States (8):
  - Central Cardiology medical Clinic, Bakersfield, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Lindner Research Center at Christ Hospital, Cincinnati, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Clinic, Danville, Pennsylvania
  - WPAHS - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Northeast Clinical Trials Group, Scranton, Pennsylvania
- Australia (3):
  - Royal North Shore Hospital, Sydney, New South Wales
  - St. George Public Hospital, Sydney, New South Wales
  - Gold Coast Hospital, Southport, Queensland
- Medical University of Vienna, Vienna, Austria
- CHR de la Citadelle, Liège, Belgium
- Brazil (7):
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Santa Isabel, Blumenau, Santa Catarina
  - Santa Casa de Marilia, Marília, São Paulo
  - Fundação Faculdade de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Mae de Deus, Porto Elegre
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
- Canada (15):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Heart Institute, Victoria, British Columbia
  - Royal Columbian Hospital, Westminster, British Columbia
  - Queen Elizabeth II Health Sciences, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - York PCI Group - Southlake Regional, Newmarket, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CSSS de Chicoutimi, Chicoutimi, Quebec
  - MUHC Royal Victoria Hospital, Montreal, Quebec
  - Quebec Heart Lung Insitute, Québec, Quebec
- China (4):
  - Shanghai Gongli Hospital, Shanghai
  - The First People's Hospital, Jiatong University, Shanghai
  - The Tenth People's Hospital Tongji University, Shanghai
  - Yueyang Hospital Shanghai University of TCM, Shanghai
- Czechia (5):
  - Krasjska Nemocnice Liberec, Liberec
  - University Hospital Pilsen, Pilsen
  - University Hospital Kralovske Vinohrady, Prague
  - University Hospital Motol, Prague
  - Masaryk Hospital, Ústí nad Labem
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - Heart Center, Tampere University Hospital, Tampere
- France (5):
  - Chu Jean Minjoz, Besançon
  - CHU Albert Michallon, Grenoble
  - Hopital Bichat, Paris
  - Hopital Lariboisiere Ap-HP, Paris
  - Centre Hospitalier de Pau, Pau
- Germany (4):
  - Universitatsklinikum Bonn, Bonn
  - Elisabeth-Krankenhaus Essen, Essen
  - Clinical Association Oberallgaeu-Kempten, Immenstadt im Allgäu
  - Klinikum der Universitat Munchen, München
- Greece (2):
  - Patras University Hospital, Pátrai
  - Ahepa University Hospital, Thessaloniki
- Hungary (2):
  - Semmelweis University Heart and Vascular Center, Budapest
  - University of Szeged, Szeged
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Waikato Hospital, Hamilton, New Zealand
- Medical University Skopje, Skopje, North Macedonia
- Clinical Center of Serbia, Belgrade, Serbia
- South Korea (4):
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Chonnam National University Hospital, Gwangju
  - Kyung-Hee University Hospital, Seoul
  - Seoul Boramae Medical Center, Seoul
- Spain (8):
  - Hospital Universitari Germans Trias I Pujol, Baldona
  - Complexo Hospitalario A Coruna, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - University Hospital La Paz, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Clinico Universitario de Vigo, Vigo
- United Kingdom (12):
  - Hampshire Hospitals NHS Fuondation Trust, Basingstoke
  - Barts and The London Heart and Chest Centre, Bethnal Green
  - Frimley Park Hospital, NHS Foundation Trust, Camberley
  - Hull and East Yorkshire Hospitals, Hull
  - Kettering General Hospital, Kettering
  - Glenfield General Hospital, Leicester
  - Manchester Royal Infirmary, Manchester
  - University Hospital South Manchester, Manchester
  - Queen Elizabeth the Queen Mother Hospital, Margate
  - Sheffield Teaching Hospitals, Sheffield
  - University Hospital Southampton, Southampton
  - Musgrove Park Hospital, Taunton

REFERENCES:
- [Background] Jolly SS, Cairns J, Yusuf S, Meeks B, Shestakovska O, Thabane L, Niemela K, Steg PG, Bertrand OF, Rao SV, Avezum A, Cantor WJ, Pancholy SB, Moreno R, Gershlick A, Bhindi R, Welsh RC, Cheema AN, Lavi S, Rokoss M, Dzavik V. Design and rationale of the TOTAL trial: a randomized trial of routine aspiration ThrOmbecTomy with percutaneous coronary intervention (PCI) versus PCI ALone in patients with ST-elevation myocardial infarction undergoing primary PCI. Am Heart J. 2014 Mar;167(3):315-321.e1. doi: 10.1016/j.ahj.2013.12.002. Epub 2013 Dec 14. PMID 24576514
- [Result] Jolly SS, Cairns JA, Yusuf S, Meeks B, Pogue J, Rokoss MJ, Kedev S, Thabane L, Stankovic G, Moreno R, Gershlick A, Chowdhary S, Lavi S, Niemela K, Steg PG, Bernat I, Xu Y, Cantor WJ, Overgaard CB, Naber CK, Cheema AN, Welsh RC, Bertrand OF, Avezum A, Bhindi R, Pancholy S, Rao SV, Natarajan MK, ten Berg JM, Shestakovska O, Gao P, Widimsky P, Dzavik V; TOTAL Investigators. Randomized trial of primary PCI with or without routine manual thrombectomy. N Engl J Med. 2015 Apr 9;372(15):1389-98. doi: 10.1056/NEJMoa1415098. Epub 2015 Mar 16. PMID 25853743
- [Derived] Alkhalil M, Kuzemczak M, Zhao R, Kavvouras C, Cantor WJ, Overgaard CB, Lavi S, Sharma V, Chowdhary S, Stankovic G, Kedev S, Bernat I, Bhindi R, Sheth T, Niemela K, Jolly SS, Dzavik V. Prognostic Role of Residual Thrombus Burden Following Thrombectomy: Insights From the TOTAL Trial. Circ Cardiovasc Interv. 2022 May;15(5):e011336. doi: 10.1161/CIRCINTERVENTIONS.121.011336. Epub 2022 May 17. PMID 35580203
- [Derived] Moxham R, Dzavik V, Cairns J, Natarajan MK, Bainey KR, Akl E, Tsang MB, Lavi S, Cantor WJ, Madan M, Liu YY, Jolly SS. Association of Thrombus Aspiration With Time and Mortality Among Patients With ST-Segment Elevation Myocardial Infarction: A Post Hoc Analysis of the Randomized TOTAL Trial. JAMA Netw Open. 2021 Mar 1;4(3):e213505. doi: 10.1001/jamanetworkopen.2021.3505. PMID 33769510
- [Derived] Jolly SS, Cairns JA, Lavi S, Cantor WJ, Bernat I, Cheema AN, Moreno R, Kedev S, Stankovic G, Rao SV, Meeks B, Chowdhary S, Gao P, Sibbald M, Velianou JL, Mehta SR, Tsang M, Sheth T, Dzavik V; TOTAL Investigators. Thrombus Aspiration in Patients With High Thrombus Burden in the TOTAL Trial. J Am Coll Cardiol. 2018 Oct 2;72(14):1589-1596. doi: 10.1016/j.jacc.2018.07.047. PMID 30261959
- [Derived] Sheth TN, Kajander OA, Lavi S, Bhindi R, Cantor WJ, Cheema AN, Stankovic G, Niemela K, Natarajan MK, Shestakovska O, Tittarelli R, Meeks B, Jolly SS. Optical Coherence Tomography-Guided Percutaneous Coronary Intervention in ST-Segment-Elevation Myocardial Infarction: A Prospective Propensity-Matched Cohort of the Thrombectomy Versus Percutaneous Coronary Intervention Alone Trial. Circ Cardiovasc Interv. 2016 Apr;9(4):e003414. doi: 10.1161/CIRCINTERVENTIONS.115.003414. PMID 27056766
- [Derived] Jolly SS, Cairns JA, Yusuf S, Rokoss MJ, Gao P, Meeks B, Kedev S, Stankovic G, Moreno R, Gershlick A, Chowdhary S, Lavi S, Niemela K, Bernat I, Cantor WJ, Cheema AN, Steg PG, Welsh RC, Sheth T, Bertrand OF, Avezum A, Bhindi R, Natarajan MK, Horak D, Leung RC, Kassam S, Rao SV, El-Omar M, Mehta SR, Velianou JL, Pancholy S, Dzavik V; TOTAL Investigators. Outcomes after thrombus aspiration for ST elevation myocardial infarction: 1-year follow-up of the prospective randomised TOTAL trial. Lancet. 2016 Jan 9;387(10014):127-35. doi: 10.1016/S0140-6736(15)00448-1. Epub 2015 Oct 22. PMID 26474811
- [Derived] Jolly SS, Cairns JA, Yusuf S, Meeks B, Gao P, Hart RG, Kedev S, Stankovic G, Moreno R, Horak D, Kassam S, Rokoss MJ, Leung RC, El-Omar M, Romppanen HO, Alazzoni A, Alak A, Fung A, Alexopoulos D, Schwalm JD, Valettas N, Dzavik V; TOTAL Investigators. Stroke in the TOTAL trial: a randomized trial of routine thrombectomy vs. percutaneous coronary intervention alone in ST elevation myocardial infarction. Eur Heart J. 2015 Sep 14;36(35):2364-72. doi: 10.1093/eurheartj/ehv296. Epub 2015 Jun 29. PMID 26129947
- [Derived] Williams PD, Mamas MA, Fraser DG. A coronary artery cast. Can J Cardiol. 2011 Nov-Dec;27(6):871.e5-6. doi: 10.1016/j.cjca.2011.08.108. Epub 2011 Oct 14. No abstract available. PMID 22000582
- See also: TOTAL - A Randomized Trial of Routine Aspiration Thrombectomy with Percutaneous Coronary Intervention (PCI) vs. PCI Alone in Patients with STEMI Undergoing Primary PCI (Population Health Research Institute) — http://www.phri.ca/